CLINICAL TRIAL: NCT07184801
Title: A Randomized Controlled Trial for Studying the Efficacy and Safety of Dexmedetomidine Vs Midazolam for Procedural Sedation During Medical Thoracoscopy
Brief Title: Safety and Efficacy of Dexmedetomidate vs. Midazolam for Procedural Sedation During Medical Thoracoscopy
Acronym: DEMISE-MT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IEC-INT/2025/DM-2480
Record Dates: First submitted 2025-09-13; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Medical Thoracoscopy
Keywords: Thoracoscopy, Midazolam, sedation
MeSH Terms: interventions — Dexmedetomidine; Midazolam; GOLPH3 protein, human

STUDY DESIGN:
Intervention Model Description: To compare the efficacy and safety of Dexmedetomidine vs Midazolam for conscious sedation among patients undergoing medical thoracoscopy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Immediately before procedure
  * 2 mL normal saline bolus
  * 1 µg /Kg fentanyl in 0.9% normal saline (10 mL dose volume) IV as slow bolus
  * Dexmedetomidine 1 µg /Kg in 0.9% normal saline (100 mL) over 10 minutes
  During entire procedure
  • Dexmedetomidine (30 mcg in 0.9% saline, 50 ml) infused at a rate of 0.5 µg /Kg/hour
  Rescue boluses
  * 0.5 µg /Kg of Fentanyl IV boluses up to 100 µg total.
  * If further need of analgesia despite 100 µg of Fentanyl, Injection Tramadol 50 mg IV bolus as needed upto 200 mg total dose.
  Interventions: Drug: Dexmedetomidine
- Group 2 (Active Comparator): Immediately before procedure
  * 2 mg midazolam
  * 1 µg /Kg Fentanyl, in 0.9% saline IV slow bolus
  * 100 mL 0.9% normal saline (100 mL) over 10 minutes During entire procedure
  * 0.9% normal saline 50 mL infused at a rate of 0.5 µg /Kg/Hr Rescue boluses
  * 0.5 µg /Kg of Fentanyl IV boluses up to 100 µg total.
  * If further need of analgesia despite 100 µg of Fentanyl, Injection Tramadol 50 mg IV bolus as needed upto 200 mg total dose.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — The patient will receive dexmedetomidine bolus dose of 1 µg /Kg over 10 minutes followed by 0.5 µg /kg/hr infusion titrated to desired sedation level (RSS 3). For patients who do not achieve an RSS of 3, we will give 1 mg bolus of midazolam. All additional boluses will be recorded. The patient will initially receive a bolus of 2 mL 0.9% normal saline intravenously for blinding purpose
  Other Names: Dexmed
  Arms: Group 1
Drug: Midazolam — The patient will receive midazolam bolus dose of 2 mg IV. They will receive an infusion of normal saline over 10 minutes for blinding purpose. Further need of sedation (as assessed by RSS) will be met by additional IV boluses of 1 mg midazolam. During the procedure they will receive continuous infusion of normal saline at a rate of 0.5 µg /Kg/Hr as placebo.
  Other Names: Midas
  Arms: Group 2

SUMMARY:
Medical thoracoscopy can be performed under procedural sedation (conscious sedation) in most of the cases. Procedural sedation is a state where the patient lies comfortably without much movement, does not feel pain and has a dissociative state (separation of mind and body. In view of the existing literature, we hypothesize that use of dexmedetomidine for procedural sedation during medical thoracoscopy will improve the ease of performing the procedure, lower the consumption of rescue analgesics and risk of intra- and post-procedure complications, improve the yield, shorten the recovery period and reduce the post-procedure pain in comparison to midazolam. In this study we propose to show that procedural sedation with dexmedetomidine during medical thoracoscopy is more beneficial for both patient and the clinician in terms of yield and shorter procedure time in comparison with conventional midazolam-fentanyl combination.

DETAILED DESCRIPTION:
Francis Richard Cruise was probably the first person to ever implement the idea of peeking into the pleural cavity with an endoscope, which he did back in 1865-1866 for examining an 11-year-old girl with tuberculous pleural effusion complicated by a pleurocutaneous fistula. However, Hans-Christian Jacobaeus was the first respiratory physician to meticulously explore the scope of diagnostic and therapeutic thoracoscopy and document it extensively as early as 1910(1). Medical thoracoscopy, so called because of the ability of the physicians to perform it under simple analgesia and conscious sedation without the need of intubation or general anaesthesia (as opposed to VATS), has come a long way since then and is currently one of the most important invasive diagnostic procedures performed by the respiratory physicians for diagnosis of pleural diseases. Mainly lauded for its high diagnostic accuracy for malignant pleural effusion (sensitivity of 97%) and pleural tuberculosis (99%)(2) after all other investigations have failed, medical thoracoscopy can also be used to evaluate and manage parapneumoic effusions, recurrent pneumothoraxes(3, 4), mediastinal disorders, diffuse lung diseases(5-7) and to perform therapeutic procedures such as adhesiolysis and pleurodesis (talc powdrage).

Medical thoracoscopy can be performed under procedural sedation (conscious sedation) in most of the cases. Procedural sedation is a state where the patient lies comfortably without much movement, does not feel pain and has a dissociative state (separation of mind and body)(8)8. Conscious sedation is preferred in this procedure because it can then be performed outside an operation theatre, and a continuous communication with the patients can be maintained. Proper level of conscious sedation is of paramount importance to perform the procedure swiftly and obtain the intended samples. British thoracic society recommends use of local anaesthesia with 1 or 2% lignocaine for local infiltration in conjunction with a benzodiazepine (midazolam) as sedative and an opioid (fentanyl) as analgesic. They point out that propofol may be an alternative in selected cases, but its administration requires presence of an anaesthesiologist(9). The NCCP-ICS joint consensus based clinical guideline on medical thoracoscopy also recommends the midazolam and fentanyl as a combination for procedural sedation(10). A survey of Indian practices on thoracoscopy found that 54.5% proceduralists use a combination of midazolam and fentanyl for procedural sedation and 1-7% use propofol or other agents in combination. Only 2% have used dexmedetomidine for this purpose(11). Although midazolam has been widely used for this purpose due to its quick onset and short duration of action, overall safety and availability of specific antidote, it is not without limitations. Midazolam does not have analgesic property and requires another opioid to be administered to relieve pain during the procedure. Boluses of midazolam are known to cause hypotensive episodes which may complicate the procedure. A recent study of gastrointestinal endoscopy also found hypoxia and failure of sedation as major adverse events associated with midazolam-induced procedural sedation(12). Dexmedetomidine, the active dextro-isomer of medetomidine, was first approved for short-term sedation in the ICU (<24 hours) in 1999. It has since gained prominence as an excellent agent for procedural sedation. It is a highly selective alpha-2 agonist (8 times the affinity of clonidine towards alpha2 receptor). It acts both pre- and post-synaptically, mainly on alpha2A-AR and alpha2C-AR isotypes. Its sedative properties are attributed to high concentration of these receptors in locus caeruleus of brainstem and the analgesic property is probably due to its action at the level of spinal cord (inhibitory action on nociceptive receptors in substantia gelatinosa of the dorsal horn). Dexmedetomidine has additional axiolytic properties. Its sympatholytic and vagomimetic actions are responsible for drop in heart rate and blood pressure, which make it an excellent agent in patients with tachycardia or hypertension. It has a distribution half-life of just 5 minutes, a plasma half-life of 2-2.5 hours and an elimination half-life of 2 hours, all of which translates into its faster onset of action and faster recovery from sedative effects. Its major side effects included hypotension and bradycardia, both of which could be promptly managed with ephedrine and atropine, respectively(13). Some studies have shown it to have some anti-inflammatory and bacterial clearance properties superior to GABA-agonists like benzodiazepines or propofol expected to improve clinical outcomes in ventilated patients with sepsis, although clinical trials failed to show any statistically significant difference in outcome measures(14-17). Moreover, there is a growing body of evidence that dexmedetomidine may reduce the risk of delirium in ICU, which has been a problem with currently used benzodiazepines like delirium. A 2019 meta-analysis (including 25 eligible papers) found that, in comparison to placebo, dexmedetomidine reduces the incidence of delirium (7.6% in dexmedetomidine group vs 18.5% in placebo group, OR 0.36, CI-95%, P<0.001) in ICU patients. This was concluded from 8 randomized clinical trials with low level of heterogeneity. 4 RCTs also pointed towards a lower level of agitation among patients receiving dexmedetomidine in comparison to placebo(18). Taking all this into consideration it appears logically sound to hypothesize that dexmedetomidine may be a better agent for procedural sedation in comparison to midazolam. A systematic review in 2017 found that dexmedetomidine sedation was associated with higher clinician and patient comfort and a higher degree of analgesia and sedation in comparison to midazolam(19). Among the procedures included in this meta-analysis, bronchoscopy was the most frequent (one study by Liao et al; n=198). Other procedures included dental and ophthalmological interventions and endoscopies. A 2021 randomized clinical trial performed in PGIMER, Chandigarh found that dexmedetomidine reduces the need of rescue sedation during EBUS-TBNA and allows for a faster post-procedure recovery albeit at the expense of slightly higher risk of hypotension and bradycardia(20). However, medical thoracoscopy should not be equated with bronchoscopy as it requires incision and insertion of the endoscope in an otherwise sterile cavity. It is associated with considerably higher degree of pain and discomfort. Henceforth the observations of this study may not be applicable in cases of medical thoracoscopy. There is very little body of evidence for comparison of dexmedetomidine and midazolam for procedural sedation in medical thoracoscopy. In 2021, a randomized clinical trial aimed at comparing midazolam-fentanyl with dexmedetomidine for procedural sedation during pluroscopy showed that although use of dexmedetomidine did not improve PF ratio during the procedure, it did have a significant advantage over midazolam-fentanyl in terms of smaller decrease in FEV1 after procedure, smaller consumption of rescue analgesics and accelerated recovery from sedation after completion of the procedure(21). A pilot RCT was done in 2022 that compared dexmedetomidine infusion and midazolam bolus for procedural sedation during medical thoracoscopy. They found that pulmonologist-rated procedural satisfaction VAS score was significantly higher and pulmonologist-rated cough VAS score, and patient-rated faces pain scale score were significantly lower in dexmedetomidine group in comparison to midazolam group. The patients in dexmedetomidine group also required lower dose of rescue analgesia(22). The problem with the study was that it had the clinicians' comfort as its primary outcome and used VAS score to compare it. The minimum clinically significant difference in VAS score is not known or validated, and hence question remains about the difference in comfort the proceduralist felt.

In view of the existing literature that has been laid out above, we hypothesize that use of dexmedetomidine for procedural sedation during medical thoracoscopy will improve the ease of performing the procedure, lower the consumption of rescue analgesics and risk of intra- and post-procedure complications, improve the yield, shorten the recovery period and reduce the post-procedure pain in comparison to midazolam. In this study we propose to show that procedural sedation with dexmedetomidine during medical thoracoscopy is more beneficial for both patient and the clinician in terms of yield and shorter procedure time in comparison with conventional midazolam-fentanyl combination.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 and ≤80 years
2. Medical thoracoscopy performed for the work-up of undiagnosed pleural effusion

Exclusion Criteria:

1. Patients with ICD in situ for more than 5 days
2. SP02<92%
3. Haemodynamic instability (systolic blood pressure ≤90 mmHg or >180mmHg, or diastolic BP >110mmHg) before the procedure
4. MI/unstable angina in the last 3 months
5. Hb<8g/dL, platelet<50000 cells/dL
6. Lack of pleural space due to adhesion
7. Uncorrected coagulopathy (PT>3 secs above control; APTT>10 secs above control
8. Failure to provide informed consent
9. Patients with known allergy or previously recorded severe adverse events to the sedatives used in the study
10. Patients who required any anaesthetic/analgesic agent in past 7 days
11. Patients on psychotropic drugs that may alter sensorium

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total amount of rescue medication (sedation or analgesia) required during MT. | 6 hours
  The total amount of rescue medication bolus will be counted

SECONDARY OUTCOMES:
Pulmonologist rated ease of the procedure (satisfaction visual analogue scale [VAS]) | 6 hours
  Operator rated ease of procedure will be analysed using VAS (0 mm being very easy; 100 being most difficult)
Pulmonologist rated incidence of cough on 100 mm VAS (cough VAS); | 6 hours
  Operator s assessment of cough during procedure will be assessed using VAS
Patient rated VAS 2 hours after completion of the procedure | 6 hours
  Patients comfort during procedure will be assessed after procedure using VAS (0 mm being very comfortable; 100 mm being very uncomfortable)
Willingness to undergo repeat thoracoscopy if required | 6 hours
  Patient's willingness to undergo procedure will be assessed using visual analogue scale (0 mm being least willing; 100 being most willing)
Adverse events | 6 hours
  intra-operative adverse effects arising because of the use of either sedative agent (midazolam+fentanyl or dexmedetomidine+fentanyl) including transient or persistent hypotension (MAP<65 for >15 minutes/requiring interventions like fluid bolus/inotrope/abandonment of procedure), bradycardia, hypoxia (Sp02<90% for >30 seconds), excessive bleeding or neurological symptoms (seizure)
Time to recovery | 6 hours
  time to achieve a score of 9 on the modified Aldrete scale
Post procedure complications | 6 hours
  Post-operative complication of the procedure following the procedure (including pain, non-expansion of lung, persistent air-leak, persistent hypoxia, persistent hypotension, haemothorax and others)

CONTACTS AND LOCATIONS:
Overall Officials: Inderpaul S Sehgal, DM, Principal Investigator — PGIMER, Chandigarh
Locations (1):
- Bronchoscopy suite, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared after reasonable request to the PI. Data will be shared only for academic purposes